CLINICAL TRIAL: NCT01721486
Title: Efficacy of IV vs Oral Administration of Acetaminophen for Pain Control Following Tonsillectomy With or Without Adenoidectomy
Brief Title: Acetaminophen's Efficacy For Post-operative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaveh Aslani, MD (Other)
Responsible Party: Sponsor-Investigator, Kaveh Aslani, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-162
Record Dates: First submitted 2012-09-27; First posted 2012-11-05 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Tonsillitis; Airway Obstruction; Difficulty Swallowing
Keywords: tonsillitis; recurrent tonsillitis; obstructed air passages; swallowing difficulties
MeSH Terms: conditions — Tonsillitis; Airway Obstruction; Deglutition Disorders | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Group (Experimental): IV acetaminophen 15 mg/kg (up to 1000 mg) administered intraoperatively over a 15 minute infusion.
  Interventions: Drug: IV acetaminophen
- Control Group (Active Comparator): PO acetaminophen elixir 15 mg/kg (up to 1000 mg) administered approximately 90 minutes (+/- 30 minutes) prior to induction of anesthesia in the pre-operative area.
  Interventions: Drug: PO acetaminophen

INTERVENTIONS:
Drug: IV acetaminophen — IV acetaminophen 15 mg/kg (up to 1000 mg) over 15 minute infusion after IV placement in OR .
  Other Names: Ofirmev
  Arms: Study Group
Drug: PO acetaminophen — PO acetaminophen elixir 15 mg/kg (up to 1000 mg) administered approximately 90 minutes (+/- 30minutes) prior to induction of anesthesia in the pre-operative area.
  Other Names: Acetaminophen Elixir
  Arms: Control Group

SUMMARY:
The purpose of this study is to compare IV acetaminophen to oral acetaminophen for pain control in children undergoing tonsillectomy with or without adenoidectomy.

DETAILED DESCRIPTION:
Tonsillectomy with or without adenoidectomy is a common surgical procedure in children and adolescents. Usually performed for recurrent tonsillitis or symptoms of airway obstruction, the procedure can result in significant post-operative pain. Common analgesic techniques include the use of oral acetaminophen, non-steroidal anti-inflammatory drugs (NSAIDs), such as ibuprofen by mouth (PO) or ketorolac intravenous (IV), and narcotics. Acetaminophen has been shown to be effective in reducing pain and post-operative opioid requirements. Its administration can be oral, rectal, or intravenous. NSAIDs, though effective for pain control, have been shown to increase bleeding risk and disrupt hemostasis. Narcotics are effective for pain control but increase the risk of nausea and vomiting. They also have the potential to cause respiratory depression.

IV acetaminophen (OFIRMEV) is indicated for management of mild to moderate pain, and as an adjunct to opioids for severe pain. Several studies have examined the efficacy of IV acetaminophen vs placebo and/or active controls (meperidine, rectal acetaminophen (PR), tramadol). IV acetaminophen has been shown to be superior to placebo for pain control. Though there is data regarding peak plasma and Cerebral Spinal Fluid (CSF) concentration of acetaminophen when given by different routes (PO vs IV vs PR), there is no data comparing the efficacy of oral vs IV administration for pain control post-tonsillectomy in children.

ELIGIBILITY:
Inclusion Criteria:

* Children 5-13 years of age
* Surgical procedure: tonsillectomy with or without adenoidectomy
* American Society of Anesthesiologists physical status classification 1 and 2 (patients that have either no systemic illness or mild systemic disease that is well-controlled, e.g. mild asthma)

Exclusion Criteria:

* Known allergy to study medication(s)
* Known genetic abnormality
* Known hepatitis
* Children with other physical, mental or medical conditions which, in the opinion of the PI, make study participation inadvisable or impairs pain assessment
* Children who have taken any analgesic within 24 hours prior to surgery
* Enrollment in concurrent research study
* Pregnant patients*
* Students/trainees/staff*
* Mentally disabled/cognitively impaired*

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kaveh Aslani, MD, Principal Investigator — Corewell Health East
Locations (1):
- Beaumont Health System, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled over a period of 23 months in the pre-operative setting of an out-patient surgical unit.
Groups:
- Study Group: IV acetaminophen 15 mg/kg (up to 1000 mg) administered intraoperatively over a 15 minute infusion.
  IV acetaminophen: IV acetaminophen 15 mg/kg (up to 1000 mg) over 15 minute infusion after IV placement in OR in study group only.
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 21 | 20
Completed | 20 | 19
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline participant number does not include 2 patients removed from study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 19 | 39
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Total Pain Medication
Description: All pain medication documented during the first 24 hours postoperatively, in mg morphine equivalents.
Time Frame: From time of PACU admission until 24 hours post-operatively.
Population: Only patients receiving rescue pain medication were analyzed.
Measure: Median (Inter-Quartile Range); unit: mg
Groups:
- Study Group: IV acetaminophen 15 mg/kg (up to 1000 mg) administered intraoperatively over a 15 minute infusion after IV placement in OR in study group only.
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 14 | 14
mg | 1.7 [0 to 5.5] | 2.2 [0 to 4.5]

2. Secondary Outcome: FLACC: Face, Legs, Activity, Cry & Consolability (FLACC) Pain Assessment Scores
Description: FLACC: Face, Legs, Activity, Cry, and Consolability Pain Assessment Scale (FLACC), a five-item, three point scale that measures each of 5 pain behaviors on a scale of 0 - 2 which are summed to result in a total score of 0 - 10. Clinical judgment is used to interpret pain. The higher the score on the FLACC correlates with a higher pain score (0= no behaviors indicative of pain and 10= five behaviors indicative of significant pain). This scale was evaluated by blinded post-operative anesthesia care unit (PACU) Registered Nurses (RNs) at admission to PACU.
Time Frame: At time of admission into PACU.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 20 | 19
units on a scale | 0 [0 to 10] | 0 [0 to 8]

3. Secondary Outcome: Incidence of Post-operative Vomiting
Description: Percentage of subjects with at least one episode of post-operative vomiting
Time Frame: From admission into PACU until 24 hours post-hospital discharge. At the conclusion of enrollment, this measure will be assessed for all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 20 | 19
Participants | 1 | 3

4. Secondary Outcome: Parental Satisfaction With Pain Control.
Description: Parental satisfaction with pain control, as measured on a 10 point Likert scale where 1= Extremely dissatisfied and 10= Extremely satisfied. Data gathered through phone call to parents 24 hours post hospital discharge.
Time Frame: 24 hours post hospital discharge.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 20 | 19
units on a scale | 9 [8 to 10] | 8 [8 to 10]

ADVERSE EVENTS:
Time Frame: Adverse events were collected after informed consent was obtained until the follow-up telephone call 24 hours following hospital discharge.
Arm/Group | Study Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/19
Other Adverse Events (participants affected / at risk) | 4/20 | 6/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Group (N=20) | Control Group (N=19)
bleeding (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=20) | Control Group (N=19)
nausea (Nervous system disorders) | 0 (0) | 1 (1)
vomit x1 (Gastrointestinal disorders) | 1 (1) | 1 (1)
vomit x2 (Gastrointestinal disorders) | 0 (0) | 1 (1)
vomit x3 (Gastrointestinal disorders) | 0 (0) | 1 (1)
PACU delirium (Nervous system disorders) | 0 (0) | 1 (1)
poss. airway swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 0 (0)
stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The number of participants in both groups are very small. Data in pain scores outcome was skewed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes